CLINICAL TRIAL: NCT03254342
Title: Magnetic Resonance Spectroscopy and Medication Response: A Pilot Study
Brief Title: MRS and Medication Response: A Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Unable to obtain a reliable MRS signal
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alan Schatzberg, Professor, Department of Psychiatry and Behavioral Sciences, Stanford University
Other Study IDs: 28162
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Major Depressive Disorder; Major Depressive Episode; Major Depressive Disorder, Recurrent; Major Depression Mild; Major Depression Moderate; Major Depression Severe
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Major depressive disorder: There is no intervention/treatment in this study.
- Non-depressed individuals: There is no intervention/treatment in this study.

SUMMARY:
We hope to demonstrate that magnetic resonance spectroscopy can detect brain concentration levels of paroxetine (Paxil) or citalopram (Celexa) or escitalopram (Lexapro) in depressed patients.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate that it is feasible to image paroxetine (Paxil) or citalopram (Celexa) or escitalopram (Lexapro) brain concentrations using MRS technology in depressed patients.

The longer-term goal is to determine the relationship between clinically administered doses of paroxetine (Paxil) or citalopram (Celexa) or escitalopram (Lexapro) (antidepressants), the amount of drug in the body via blood level, the concentrations of the drug achieved in brain measured via MRS, and genetics.

It has been previously reported that individuals taking 20mg of paroxetine daily had brain paroxetine [(Paxil) levels via MRS ranging from 2-13 micromolar. Similar or slightly higher ranges of brain drug concentrations have been reported for fluoxetine and fluvoxamine.

Since not all depressed patients respond to medications, one reason may be the amount of medication that crosses the blood-brain barrier. This may be influenced by genetic information. We want to examine these issues on a larger scale, but first we need to demonstrate that we can indeed determine paroxetine [(Paxil) or citalopram (Celexa) or escitalopram (Lexapro)] levels via MRS.

Intended results analysis could not be conducted because a reliably sensitive spectroscopic method could not be developed.

ELIGIBILITY:
Major depressive disorder:

Inclusion Criteria:

1. DSM diagnosis of Major Depressive Disorder
2. Taking paroxetine [(Paxil) or citalopram (Celexa) or escitalopram (Lexapro)]for at least 6 weeks
3. Between 21 - 75 years of age.
4. Taking a stable dose of paroxetine [(Paxil) or citalopram (Celexa) or escitalopram (Lexapro)] for at least the 2 weeks prior to the imaging session

Healthy controls:

1. Between 21 - 75 years of age.
2. Have a 21-item HAM-D score of less than or equal to 5.
3. No current, or history of any Axis I disorder.

Identify exclusion criteria.

Exclusion criteria are as follows:

1. Contraindications for an MRI exam. These includes biomedical devices such as pacemakers, aneurysm clips, prostheses, and other metallic objects embedded in the body such as bullets, buckshot, shrapnel, and any metal fragments from working around metal.
2. Current pregnancy or lactation.
3. Patients with claustrophobia.
4. History, or current Axis I or Axis II disorders
5. Active unstable medical problems, as confirmed by screening procedures
6. Diagnosed with any autoimmune disease, (e.g., rheumatoid arthritis, Lupus, MLS).
7. Chronic use of steroids or opiates.
8. Positive urine toxicology screen for illicit substances of abuse.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Psychiatry clinic; local community.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-08-06 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Measurement of paroxetine (Paxil), citalopram (Celexa) or escitalopram (Lexapro) brain concentrations. | Within 7 Days following MRS
  Measurement of paroxetine (Paxil), citalopram (Celexa) or escitalopram (Lexapro) brain concentrations using MRS technology in depressed participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Psychiatry and Biobehavioral Sciences, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Currently there is no plan.
Supporting Information: Study Protocol, ICF